CLINICAL TRIAL: NCT04919239
Title: Double-Blind, Randomized, Placebo-Controlled, Phase IIb Clinical Trial to Investigate the Efficacy of RUTI® Therapeutic Vaccination as Adjuvant of Tuberculosis Chemotherapy
Brief Title: Clinical Trial to Investigate Therapeutic Vaccine (RUTI) Against Tuberculosis (TB)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Archivel Farma S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RUTIP2-2019-01
Record Dates: First submitted 2021-05-31; First posted 2021-06-09 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Tuberculosis, Pulmonary
MeSH Terms: conditions — Tuberculosis, Pulmonary

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RUTI® arm (Experimental): A dose of 25 μg of of RUTI vaccine will be given at week 1 (Cohort A-DS TB Patients) or month 1 (Cohort B-MDR TB Patients) after starting standard TB treatment.
  Interventions: Biological: RUTI®
- Placebo arm (Placebo Comparator): Placebo will be given at week 1 (Cohort A-DS TB Patients) or month 1 (Cohort B-MDR TB Patients) after starting standard TB treatment.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: RUTI® — Participants randomised to this arm will receive one single dose of RUTI® vaccine in the right/left deltoid muscle.
  Arms: RUTI® arm
Biological: Placebo — Participants randomised to this arm will receive aone single dose of matching RUTI® placebo in the right / left deltoid muscle.
  Arms: Placebo arm

SUMMARY:
Prospective, randomized, double-blind, multicentre, placebo-controlled clinical phase IIb trial to evaluate efficacy of RUTI® vaccine in DS- (Drug-Sensitive) and MDR-TB (Multidrug-resistant) patients favourably responding to standard MDR-TB treatment. Time point of vaccination starts upon completion of 1 week of standard DS-TB treatment (cohort A), and another cohort of patients will be vaccinated upon completion of 1 month of standard MDR-TB treatment (cohort B). All the patients will be followed up to the end of the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with pulmonary DS- or MDR-TB, and managed with standard-care TB drugs accordingly;
2. Attending a TB unit / hospital routinely diagnosed with pulmonary DS- or MDR-TB with clinical status ≥ 6 with Bandim TB score combined with chest radiography; and microbiological criteria (MGIT sputum culture), by using rapid genetic testing, gene Xpert;
3. Patients who have not received any anti-tubercular treatment in last 6 months
4. Females and males aged ≥ 18;

   * females of non-childbearing potential: at least 2 years post- menopausal or surgically sterile (e.g. tubal ligation);
   * females of childbearing potential (including females less than 2 years postmenopausal) must have a negative pregnancy test at enrolment and must agree to use highly effective methods of birth control (i.e. diaphragm plus spermicide or male condom plus spermicide, oral contraceptive in combination with a second method, contraceptive implant, injectable contraceptive, indwelling intrauterine device, sexual abstinence, or a vasectomized partner) while participating in the study;
   * males must agree to use a double barrier method of contraception (condom plus spermicide or diaphragm plus spermicide) while participating in the study; or the male patient or his female partner must be surgically sterile (e.g. vasectomy, tubal ligation) or the female partner must be post-menopausal;
5. The patient must provide written informed consent;
6. The patient must be willing and able to attend all study visits and comply with all study procedures.

Inclusion criteria for vaccination

1. Having successfully completed 1 week or 1 month (depending on the cohort) of DS or MDR-TB treatment, respectively, fully supervised; and with beneficial initial response to therapy, evidenced by clinical response.

Exclusion Criteria:

1. Inability to provide written informed consent;
2. Women reported, or detected, or willing to be pregnant during the trial period;
3. Severity of illness precluding full evaluation: expected early death, evidenced by respiratory failure, low blood pressure, WHO performance score 3-4
4. Patients with extra-pulmonary tuberculosis
5. Major co-morbid conditions precluding full evaluation, i.e., HIV positive, chronic renal failure, chronic liver failure, Malignancy, patients taking any immunosuppressant drug, active lung cancer, acute coronary syndrome, heart failure exceeding NYHA class 2;
6. Presence of secondary immunodeficiency states: Organ transplantation, diabetes mellitus
7. Any of the following laboratory parameters:

   * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3 x upper limit of normal (ULN)
   * Total bilirubin > 2 x ULN
   * Neutrophil count ≤ 500 neutrophils / mm3
   * Platelet count < 50,000 cells / mm3
8. Cytotoxic chemotherapy or radiation therapy within the previous 3 months;
9. Blood transfusion in the last three weeks prior to the trial; 10.Patients with history of alcohol or drug abuse

11. Documented allergy to TB vaccines, notably, to the RUTI® vaccine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2021-09-22 (Actual); Primary Completion 2025-06-19 (Actual); Study Completion 2025-06-19 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with Sputum Culture Negative | Up to Week 2 for Cohort A and Month 1.5 for Cohort B
  Difference between intervention and control group

SECONDARY OUTCOMES:
Percentage of patients with Sputum Culture Negative | Up to Week 8 for Cohort A and Month 6 for Cohort B
  Difference between intervention and control group
Proportion of patients with reduction of bacillary load | Up to Week 2 and 8 (Cohort A); and Months 1.5 and 6 (Cohort B)
  Difference between intervention and control group based upon Time to detection (TTD) signal in MGIT
Proportion of patients with improvement of clinical signs and symptoms | Up to Week 2 and 8 (Cohort A); and Months 1.5 and 6 (Cohort B)
  Difference between intervention and control group based upon Bandin

OTHER OUTCOMES:
Clinical safety parameters related to vaccination | Through study completion, an average of 2 year
  Serious adverse events (SAEs) by CTCAE v4.0
Local tolerability | Up to Week 8
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 in terms of site of injection for redness, pain, swelling, induration and functional limitation

CONTACTS AND LOCATIONS:
Overall Officials: Randeep Guleria, Prof, Principal Investigator — All India Institute of Medical Sciences
Locations (2):
- India (2):
  - All India Institute of Medical Sciences (AIIMS), New Delhi
  - Agartala Government Medical College (AGMC), Tripura

IPD SHARING:
Plan to Share IPD: Undecided